CLINICAL TRIAL: NCT04118699
Title: Efficacy and Safety of Rifaximin for Patients With Chronic Intestinal Pseudo-obstruction: a Single Center, Randomized, Placebo Controlled, Double-blind Phase 2 Trial
Brief Title: Efficacy and Safety of Rifaximin for Patients With Chronic Intestinal Pseudo-obstruction: a Phase 2 Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yokohama City University (Other)
Collaborators: ASKA Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YCU19001
Record Dates: First submitted 2019-09-23; First posted 2019-10-08 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Chronic Intestinal Pseudo-obstruction
Keywords: Rifaximin; L-105; phase 2 trial; CIPO; small intestinal bacterial overgrowth; systemic scleroderma
MeSH Terms: conditions — Intestinal Pseudo-Obstruction; Scleroderma, Systemic | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Experimental): Two tablets of the investigational product per dosing (400 mg of rifaximin) are orally administered 3 times daily for 4 weeks.
  Interventions: Drug: Rifaximin oral tablet
- Placebo (Placebo Comparator): Two tablets of the placebo are orally administered 3 times daily for 4 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Rifaximin oral tablet — Patients with chronic idiopathic intestinal pseudo-obstruction (CIIPO) or patients with chronic intestinal pseudo-obstruction (CIPO), secondary to systemic scleroderma, are administered investigational product (rifaximin) for 4 weeks
  Other Names: L-105
  Arms: Rifaximin
Drug: Placebo oral tablet — Patients with chronic idiopathic intestinal pseudo-obstruction (CIIPO) or patients with chronic intestinal pseudo-obstruction (CIPO), secondary to systemic scleroderma, are administered placebo for 4 weeks
  Arms: Placebo

SUMMARY:
The objective of the study is to investigate efficacy and safety of rifaximin (L-105) in patients with chronic idiopathic intestinal pseudo-obstruction(CIIPO) or patients with chronic intestinal pseudo-obstruction (CIPO), secondary to systemic scleroderma

DETAILED DESCRIPTION:
This is a placebo-controlled, randomized, double-blind, parallel group, comparative study, when patients with chronic idiopathic intestinal pseudo-obstruction(CIIPO) or patients with chronic intestinal pseudo-obstruction (CIPO), secondary to the onset of systemic scleroderma, are administered rifaximin at 400 mg 3 times daily for 4 weeks. In addition, the time course of symptoms of the patients are to be confirmed for 8 weeks after the end of administration.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged ≥20 and <75 on the day of informed consent (IC)
* Patients with CIIPO (designated intractable disease 99) at enrollment, satisfying all the criteria specified in (1) to (7) of the CIIPO Diagnostic Criteria issued in 2014 by the MHLW Research Group, or patients with CIPO, secondary to systemic scleroderma, satisfying all the same criteria specified in (1) to (6)
* Patients' levels of abdominal bloating symptoms, 4 scales of GSS, should be score 2 or 3 at the time of IC acquisition and enrollment.

Exclusion Criteria:

* Patients with malignant diseases (excluding those whose symptoms are stable and who do not require aggressive treatments such as chemotherapy and/or surgical therapy)
* Patients with psychiatric diseases (excluding those whose symptoms are stable, and the investigator or coinvestigator concludes that efficacy of the patient can be assessed without any issue)
* Patients with severe diabetes within 5 weeks before enrollment (HbA1c >10%)
* Patients who have already had gastrostomy (including percutaneousendoscopic gastro -jejunostomy, PEG-J), enterostomy, or colostomy
* Patients who underwent intestinal decompression therapy not associated with surgical procedures (trans-nasal ileus tube) within 4weeks before enrollment
* Patients who used antimicrobials, antiparasitics or antifungals (excluding topical use) within 4 weeks before enrollment
* Patients who have changed the doses of the following concomitantly administered drugs within 4 weeks before enrollment: mosapride, daikenchuto, metoclopramide, acotiamide
* Patients with severe hepatic disorders within 5 weeks before enrollment (who meet either one of the following criteria: AST≥ 5 x the upper limit of the common reference value specified in the Japanese Committee for Clinical Laboratory Standards (JCCLS), ALT≥ 5 x the upper limit of the common reference value specified in JCCLS, total bilirubin ≥ 3 x the upper limit of the common reference value specified in JCCLS, decompensated hematic cirrhosis, or jaundice)
* Patients who are pregnant, breastfeeding, possibly pregnant, or those who wish to become pregnant
* Patients with a previous history of hypersensitivity to any investigational product ingredients
* Patients with active tuberculosis
* Patients who participated in other clinical trial (including a trial with an investigational product) within 12 weeks before this enrollment and who received an intervention with a test drug
* Other patients whose participation in the trial is concluded to be inappropriate by the investigator or coinvestigator

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Improvement ratio (%) in abdominal bloating score in Global Symptomatic Score (GSS) | at the end of administration (4 weeks)
  Abdominal bloating score in Global Symptomatic Score (GSS) is used. GSS is a 4-point Likert scale ranging from 0 (no symptom) to 3 (severe, incapacitating with inability to perform normal activities), with lower scores reflecting better symptoms. Score 0 or 1 is defined as improvement.
Improvement ratio (%) in Gastrointestinal (GI) symptoms score | at the end of administration (4 weeks)
  Gastrointestinal score (GI score) is a 5-point Likert scale (0; greatly improved, 1; improved, 2; no change, 3; worsened, 4; severely worsened), with lower scores reflecting more improved symptoms. Score 0 or 1 is defined as improvement.

SECONDARY OUTCOMES:
Changes of the improvement ratio (%) in abdominal bloating score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Abdominal bloating score in Global Symptomatic Score (GSS) is used. GSS is a 4-point likert scale ranging from 0 (no symptom) to 3 (severe, incapacitating with inability to perform normal activities), with lower scores reflecting better symptoms. Score 0 or 1 is defined as improvement.
Changes of abdominal bloating score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Abdominal bloating score in Global Symptomatic Score (GSS) is used. GSS is a 4-point likert scale ranging from 0 (no symptom) to 3 (severe, incapacitating with inability to perform normal activities), with lower scores reflecting better symptoms.
Changes of the improvement ratio (%) in gastrointestinal symptoms score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Gastrointestinal score (GI score), a 5-point likert scale (0; greatly improved, 1; improved, 2; no change, 3; worsened, 4; severely worsened), with lower scores reflecting more improved symptoms, is used. Score 0 or 1 is defined as improvement.
Changes of the "good" ratio (%) in gastrointestinal symptoms score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Gastrointestinal score (GI score), 5-point likert scale (0; very good, 1; good, 2; average, 3; bad, 4; extremely bad), with lower scores reflecting better conditions, is used. Score 0 or 1 is defined as ''good''.
Changes of each score in Global Symptomatic Score other than abdominal bloating score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Global Symptomatic Score (GSS), a 4-point likert scale ranging from 0 (no symptom) to 3 (severe), of the following symptoms are assessed; (a. diarrhea, b. epigastric pain/ discomfort, c. pain in the lower quadrant/discomfort, d. tenderness, e. nausea, f. vomiting).
Changes of total scores in Global Symptomatic Score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Sum of Global Symptomatic Score (GSS) of the following 7 symptoms, 0 to maximum of 21, are assessed; (a. diarrhea, b. epigastric pain/discomfort, c. abdominal distention, d. pain in the lower quadrant/discomfort, e. tenderness, f. nausea, g. vomiting).
Changes of the improvement ratio (%) in General health condition (symptoms) score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  General health condition (symptoms) score, a 5-point likert scale (0; greatly improved, 1; improved, 2; no change, 3; worsened, 4; severely worsened), with lower scores reflecting more improved symptoms, is used. Score 0 or 1 is defined as improvement.
Changes of the "good" ratio (%) in General health condition (symptoms) score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  General health condition (symptoms) score, 5-point scale (0; very good, 1; good, 2; average, 3; bad, 4; extremely bad), with lower scores reflecting better conditions, is used. Score 0 or 1 is defined as ''good''.
Patient satisfaction score | At the end of the administration (4 weeks)
  % of the "satisfaction" ratio in patient satisfaction score
Changes of Short Form (SF)-8 health survey score | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  SF-8(short form-8), a self-reporting health survey ranging from 8 to maximum of 42, with lower scores reflecting better conditions, is used.
Small intestinal volume measured by abdominal CT scan | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Changes of small intestinal volume measured by abdominal CT scan
Changes from baseline of serum albumin level | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Serum albumin level is calculated for nutritional assessment
Changes from baseline of prealbumin (transthyretin) | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Prealbumin (transthyretin) is calculated for nutritional assessment
Changes from baseline of cholinesterase | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Cholinesterase is calculated for nutritional assessment
Changes from baseline of folic acid | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Folic acid is calculated for nutritional assessment
Changes from baseline of vitamin B12 (cobalamin) | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Vitamin B12 (cobalamin) is calculated for nutritional assessment
Changes from baseline of serum iron | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Serum iron is calculated for nutritional assessment

OTHER OUTCOMES:
Small intestinal bacterial overgrowth (SIBO) in a glucose-hydrogen breath test | Before, 4 weeks after administration;and 8 weeks after the end of administration
  Elimination rate of SIBO in a glucose-hydrogen breath test
Changes of Serum endotoxin activity | Before, 2 and 4 weeks after administration;and 4 and 8 weeks after the end of administration
  Serum endotoxin activity, ranging from 0.00-1.00, is assessed using EAA® (endotoxin activity assay, Toray Medical Co., Ltd.), FDA approved rapid whole blood assay for detection of human endotoxemia. 0.00-0.39 means low level, 0.40-0.59 means middle level, and ≥0.60 means high level.
Fecal test (intestinal flora) | Before and 4 weeks after administration
  Changes of intestinal flora detected by 16SrDNA amplicon analysis using next generation sequencing.
Adverse events | From the start of administration to 8 weeks after the end of administration
  Incidence of adverse events
Changes from baseline of hematological parameters | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Hematological parameters (red blood cell count, hematocrit, white blood cell count, platelet count) are calculated for safety assessment
Changes from the baseline of total protein | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Total protein is calculated for safety assessment
Changes from the baseline of liver function | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Liver function parameters (aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transpeptidase, alkaline phosphatase, total bilirubin) are calculated for safety assessment.
Changes from the baseline of renal function | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Creatinine and blood urea nitrogen are calculated for safety assessment.
Changes from the baseline of electrolytes | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Electrolytes (sodium, potassium, chlorine, calcium) are calculated for safety assessment.
Changes from the baseline of blood lipid level | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Blood lipid level (total cholesterol, triglyceride, and high-density lipoprotein cholesterol) is calculated for safety assessment.
Changes from the baseline of C reactive protein | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  C reactive protein is calculated for safety assessment.
Changes from the baseline of serum glucose level | Before, 2 and 4 weeks after administration; and 4 and 8 weeks after the end of administration
  Serum glucose level is calculated for safety assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Yokohama city university, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohkubo H, Iida H, Takahashi H, Yamada E, Sakai E, Higurashi T, Sekino Y, Endo H, Sakamoto Y, Inamori M, Sato H, Fujimoto K, Nakajima A. An epidemiologic survey of chronic intestinal pseudo-obstruction and evaluation of the newly proposed diagnostic criteria. Digestion. 2012;86(1):12-9. doi: 10.1159/000337528. Epub 2012 Jun 15. PMID 22710349
- [Background] Parodi A, Sessarego M, Greco A, Bazzica M, Filaci G, Setti M, Savarino E, Indiveri F, Savarino V, Ghio M. Small intestinal bacterial overgrowth in patients suffering from scleroderma: clinical effectiveness of its eradication. Am J Gastroenterol. 2008 May;103(5):1257-62. doi: 10.1111/j.1572-0241.2007.01758.x. Epub 2008 Apr 16. PMID 18422815